CLINICAL TRIAL: NCT04142151
Title: The Randomized, Double-blind, Placebo-controlled Clinical Trail of Sanchitongshu Combined Antiplatelet Drug to Prevent High-risk Ischemic Stroke Recurrence
Brief Title: Double Randomized and Placebo Controlled Trail of Sanchitongshu Combined Antiplatelet Drug to Prevent Ischemic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: XH-19-007
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-09

CONDITIONS: Ischemic Stroke; Antiplatelet Effect
Keywords: Ischemic stroke, Sanchitongshu, Aspirin, Clopidogrel
MeSH Terms: conditions — Ischemic Stroke | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SanchiTongshu group (Active Comparator): Drug: SanchiTongshu The study drugs were manufactured according to Good Manufacturing Practice (GMP) by the Pharmaceutical Factory of Chengdu Huasun Group Inc. Ltd. and presented in the form capsules. Every Sanchitongshu capsule weighed 200 mg, contained 100 mg of panaxatriol saponin (PTS) and 100 mg inactive excipient (starch). PTS comprised of dried extracts from roots of Radix Notoginseng, and had been standardised with respect to Ginsenoside Rg1 (50%), Ginsenoside Re (6%), Notoginsenoside R1 (11%). The amounts of the active ingredients were determined by analytical RP-HPLC using an acetonitrile-water gradient system as mobile hase. The peaks were detected by UV-DAD.
  Drug: Aspirin or Clopidogrel
  Interventions: Drug: Sanchitongshu; Drug: Aspirin; Drug: Clopidogrel
- SanchiTongshu Placebo group (Placebo Comparator): Drug: placebo of Sanchitongshu The Sanchitongshu placebo capsule contained dark brown muscovado sugar and the same inactive excipient (starch).
  Drug: Aspirin or Clopidogrel
  Interventions: Drug: Aspirin; Drug: Clopidogrel; Drug: placebo of Sanchitongshu

INTERVENTIONS:
Drug: Sanchitongshu — SanchiTongshu capsule produced by Chengdu Huashen Group Co., Ltd.
  Other Names: Radix/Rhizoma Notoginseng extract
  Arms: SanchiTongshu group
Drug: Aspirin — Aspirin produced by Bayer Co., Ltd.
  Other Names: Bayaspirin Enteric-coated Tablets
Drug: Clopidogrel — Clopidogrel produced by Shenzhen Salubris Co., Ltd.
  Other Names: Clopidogrel Bisulfate
Drug: placebo of Sanchitongshu — SanchiTongshu palcebo capsule contained dark brown muscovada sugar and the same inactive excipient (starch). Produced by Chengdu Huashen Group Co., Ltd.
  Other Names: Placebo
  Arms: SanchiTongshu Placebo group

SUMMARY:
This clinical trail will evaluate the effect of Sanchitongshu combined with antiplatelet drugs (Aspirin or Clopidogrel) in the treatment of high-risk ischemic stroke patients in adults. Half of participants will receive SanchiTongshu and one of antiplatelet drugs (Aspirin or Clopidogrel) in combination, while the other half will receive a placebo and one of antiplatelet drugs (Aspirin or Clopidogrel).

DETAILED DESCRIPTION:
The aim of this clinical trail is to evaluate the effect of Sanchitongshu in the treatment of high-risk ischemic stroke patients in adults. All patients included in the study should meet the inclusion criteria. All participants will receive one of antiplatelet drugs (Aspirin or Clopidogrel). Half of participants will receive Sanchitongshu and Aspirin or Clopidogrel, while the other half will receive a placebo and Aspirin or Clopidogrel. All participants will be assigned to either the active group or the control group randomly. During the clinical trail both doctors and patients are double-blind except serious adverse events occurred.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 20yrs to 85yrs;
2. Anticipated patients within 8-90 days without cardiac ischemic stroke; Responsible lesions of all cases must be confirmed by a head MRI;
3. have ability to take the drugs;
4. No serious complications, liver and kidney function is normal;
5. At least one of the following (a-c):

   1. Confirmed by MRA, CTA or DSA that stenosis of intracranial aorta beyond 50% (in A2, M2 or P2)
   2. Confirmed by MRA, CTA or DSA that stenosis of cranial artery beyond 50% (carotid artery, intra-carotid artery, vertebral artery, head artery, or lower collarbone artery)
   3. ESRS score beyond 3
6. Take Clopidogre or aspirin alone for antiplatelet treatment with informed consent
7. Willing to participate in the clinical trial and willing to be followed up with, have signed informed consent

Exclusion Criteria:

1. Younger than 20 yrs or elder than 85 yrs;
2. The neurological function defects caused by brain hemorrhage or other conditions (e.g. vascular malformations, tumors, abscesses or other non-ischemic cerebrovascular diseases);
3. Isolated sensory symptoms (e.g. numbness), isolated visual abnormalities, isolated dizziness and dizziness but have no responsibility lesions in head MRI;
4. Stroke is caused by angiography or surgery operation;
5. Stroke caused by cardio-induced embolism according to TOAST;
6. Anticoagulant evidence (heart thrombosis, such as atrial fibrillation, heart valve replacement surgery operation)
7. Contraindications of MRI examination, such as claustrophobia or implanted pacemakers
8. Severe heart and lung impairment; liver function laboratory indicator AST or ALT is 2x maximum normal value, or renal function laboratory indicator serum creatinine is 1.5X maximum normal value;
9. Plan to accept vascular surgery during the trial period (e.g. epidermal angioplasty, stent placement and bypass transplants, etc.); Surgical or interventional treatment requires discontinuation of research drugs
10. History of drug elution coronary stent implantation within one year
11. Congestive heart failure or uncontrolled Angina pectoris;
12. Platelet reduction (platelet count less than 10000/mm3);
13. Symptomatic non-traumatic intracranial bleeding, any other bleeding disorder, bleeding tendency or clotting dysfunction;
14. History of gastrointestinal ulcers, gastrointestinal bleeding, or surgical history within the last 3 months;
15. Severe complications of non-cardiovascular and life expectancy less than 3 months;
16. Have malignant tumors which in course of treatment;
17. History of allergies to SanqiTongshu;
18. Aspirin users have any of the following conditions: (1) History of allergy to aspirin or salicylic acid analogues (2) Pepsi ulcers (3) asthma or asthma history caused by aspirin;
19. Allergy history of clopidogrel;
20. History of alcohol or drugs abuse in the past 12 months;
21. Pregnant, lactating women, or women who do not take effective contraception;
22. There are other serious diseases or abnormal laboratory results who is not suitable to participate the study;
23. Those who are participating in other clinical trials or clinical trials completed in past 3 months;
24. Patients do not understand the study, or are unable to/unwilling to follow the provisions of the clinical trial.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
New stroke attack | 24 hours
  Any type of stroke events attack or recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Zhenguo Liu, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Zhenguo Liu, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided